CLINICAL TRIAL: NCT03637010
Title: Purdue Study for the Benefits of Breakfast in the Classroom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Nutrition Sciences, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1807020818
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Breakfast
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breakfast in the Classroom (Other): Baseline data will be collected to include anthropometric measures, participant characteristics, and past eating habits. For the first 8 weeks, the students will be provided with breakfast meals containing the USDA nutrition requirements. These meals are typically higher in carbohydrates and lower in protein. For the second 8 weeks, the students will be provided with higher-protein breakfast meals. These meals also contain the USDA nutrition requirements but include high-quality protein-rich foods. For the remaining 8 weeks, the students will be provided both types of meals and will be permitted to choose which they prefer to consume each day. At the end of each 8-week period, eating habits, appetite, mood, cognitive performance, and anthropometrics will be completed along with measurements of breakfast waste.
  Interventions: Other: Breakfast in the Classroom

INTERVENTIONS:
Other: Breakfast in the Classroom — For all breakfasts, the students will use the 'grab and go' approach from hallway kiosks. The students will take the breakfasts back to their respective classroom and consume them there.

SUMMARY:
This study is a 24-week crossover design study in adolescents enrolled in the 6-8th grade within the Center School District in the Kansas City, MO. This school will begin their 'Breakfast in the Classroom' program during the fall 2018 school year. Baseline data will be collected to include anthropometric measures, participant characteristics, and past eating habits. For the first 8 weeks, the students will be provided with breakfast meals containing the USDA nutrition requirements. These meals are typically higher in carbohydrates and lower in protein. For the second 8 weeks, the students will be provided with higher-protein breakfast meals. These meals also contain the USDA nutrition requirements but include high-quality protein-rich foods. For the remaining 8 weeks, the students will be provided both types of meals and will be permitted to choose which they prefer to consume each day. At the end of each 8-week period, eating habits, appetite, mood, cognitive performance, and anthropometrics will be completed along with measurements of breakfast waste.

ELIGIBILITY:
Inclusion Criteria:

* All students who are willing to participate are eligible (except Wards of the State)

Exclusion Criteria:

* Wards of the State

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Breakfast in the Classroom Participation Questionnaire | change from baseline at 8-weeks, 16 weeks, and 24-weeks.
  Questionnaires assessing whether they ate breakfast or skipped breakfast will be completed for 5 consecutive days. There are two options: yes (they did consume breakfast prior to arriving at school) or no (did not consume breakfast prior to arriving at school).

SECONDARY OUTCOMES:
Habitual Breakfast Habits Questionnaire - At School | change from baseline at 8-weeks, 16 weeks, and 24-weeks.
  During one day, a questionnaire assessing previous breakfast habits will be given to participants. This questionnaire asks how many days per week they consume various breakfast foods. There are 17 breakfast options, and they will report how many times per week they have consumed them over the past month. The options include never, 1-2 times per week, 3-4 times per week, or every school day.
Habitual Breakfast Habits Questionnaire - At Home | change from baseline at 8-weeks, 16 weeks, and 24-weeks.
  During one day, a questionnaire assessing previous breakfast habits will be given to participants. This questionnaire asks how many days per week they consume various breakfast foods. There are 17 breakfast options, and they will report how many times per week they have consumed them over the past month. The options include never, 1-2 times per week, 3-4 times per week, 5-6 times per week, or every day.
Benefits of Breakfast Questionnaire | change from baseline at 8-weeks, 16 weeks, and 24-weeks.
  During one day, a questionnaire asking the participants what happens when participants consume breakfast and skip breakfast will be administered. They will be given a list of choices (multiple selections are allowed) and the units for analysis will be binary (they chose it or did not choose it).
Snacking Questionnaires | change from baseline at 8-weeks, 16 weeks, and 24-weeks.
  During one day, questionnaires assessing typical snacking behavior will be completed once. Participants will be asked how many times they ate 18 specific foods/food groups throughout the past week. The options include none, 1 total, 2-4 total, 5-6 total, 1 each day, 2-3 each day, or 4+ each day. The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available).
Cognitive Performance Assessment | 8-weeks, 16 weeks, and 24-weeks post intervention
  During one day, cognitive performance assessments will occur once prior to lunch and after breakfast using the online CNS Vital Signs neurocognitive assessment system during one day. The CNS Vital Signs system contains a battery of computerized tests to assess attention, memory, executive function, and cognitive flexibility. The assessment will occur outside of classroom learning activities.
Hunger Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing hunger will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, and before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Fullness Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing fullness will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, and before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Prospective Food Consumption Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing prospective food consumption will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, and before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Energy Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing energy will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Sleepiness Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing sleepiness will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Happiness Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing happiness will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Stress Questionnaires | 8-weeks, 16 weeks, and 24-weeks post intervention
  Questionnaires assessing stress levels will be completed during the following times for 3 consecutive days: before breakfast, immediately after breakfast, 60 minutes after breakfast, 120 minutes after breakfast, before lunch. The questions are worded as "how strong is your feeling of" or "how strong is your desire" with anchors of "not at all" to "extremely." The students will complete these on their respective Chromebook laptops or will be provided paper copies (if their Chromebook is not available). All results will be a number from 0 ("not at all") to 100 ("extremely") with the unit "of out of 100."
Breakfast Plate Waste | 8-weeks, 16 weeks, and 24-weeks post intervention
  For 5 days, the students will be asked to place all uneaten breakfasts into labeled baggies and discard in the bins at the front of the room. Research staff will weigh the meals prior to being delivered to the hallway kiosks and will re-weight the meals once the students are finished with breakfast.
Body Mass Index Change | change from baseline at 8-weeks, 16 weeks, and 24-weeks.
  Body mass index (units of kg/m^2) will be calculated based on body weight and height of participants. Body weight will be measured to the nearest tenth of a kg using a standard scale. Height will be assessed with a stadiometer or wall ruler (to the nearest tenth of a centimeter). Both procedures will be measured in a private room.

CONTACTS AND LOCATIONS:
Locations (1):
- Center Middle School, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided